CLINICAL TRIAL: NCT00005700
Title: Fat Reduction Intervention Trial in African-Americans
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4281; R01HL051508 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2001-05

CONDITIONS: Cardiovascular Diseases; Coronary Heart Disease Risk Reduction; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To conduct a randomized controlled trial to evaluate the effectiveness of an intervention to reduce dietary fat.

DETAILED DESCRIPTION:
BACKGROUND:

The African-American population of the United States continues to experience high rates of mortality from cardiovascular (CV) disease, including coronary heart disease, stroke and renal failure. The major syndromes which determine CV risk, including obesity, hypercholesterolemia, glucose intolerance, and hypertension, all occur more frequently among African Americans. Nutritional factors underlie many forms of CV disease and are an important focus of current prevention efforts. Very little is currently known, however, about specific nutritional patterns among African Americans that might lead to CV risk, or the applicability of structured interventions.

The study was conducted in response to an initiative on "Collaborative Projects on Minority Health" which was released in October 1992 after review and approval at the September 1992 National Heart, Lung, and Blood Advisory Council.

DESIGN NARRATIVE:

Given the growing recognition of the importance of total fat, from the point of view of both disease risk and eating patterns, the primary focus of the intervention was to reduce the percentage of calories in the diet from fat. Four hundred households were recruited and randomly assigned to either an active intervention or observation group for a period of 18 months. Dietary change consistent with specific recommendations made to the American public for reducing cardiovascular (CV) risk was encouraged, namely, reduction in total fat, saturated fat (SFA), and cholesterol (Chol). A practical, community-based program was developed which could be taken into households. Nutrition education and enhancement of skills helpful in making behavioral change formed the basis of the intervention. Lay educators, recruited from the target neighborhoods, worked under the close supervision of a community nutritionist. Changes in reported dietary intake, serum lipids/lipoproteins and body weights were measured. In addition to the formal evaluation of the trial outcome, an important secondary goal was to obtain detailed information about eating patterns in this community and characterize behavior associated with the achievement and maintenance of target nutrient goals.

The study was part of a collaborative project on minority health. Dr. Prewitt collaborated with Dr. Marian Fitzgibbon who was the principal investigator on R01HL51532.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-09; Study Completion 1998-08 (Actual)

REFERENCES:
- [Background] Prewitt TE, Durazo-Arvizu R, McGee DL, Luke A, Cooper RS. One size fits all: implications for assessing dietary behavior. J Am Diet Assoc. 1997 Jul;97(7 Suppl):S70-2. doi: 10.1016/s0002-8223(97)00734-7. PMID 9216572
- [Background] Luke A, Durazo-Arvizu R, Rotimi C, Prewitt TE, Forrester T, Wilks R, Ogunbiyi OJ, Schoeller DA, McGee D, Cooper RS. Relation between body mass index and body fat in black population samples from Nigeria, Jamaica, and the United States. Am J Epidemiol. 1997 Apr 1;145(7):620-8. doi: 10.1093/oxfordjournals.aje.a009159. PMID 9098179
- [Background] Fitzgibbon ML, Prewitt TE, Blackman LR, Simon P, Luke A, Keys LC, Avellone ME, Singh V. Quantitative assessment of recruitment efforts for prevention trials in two diverse black populations. Prev Med. 1998 Nov-Dec;27(6):838-45. doi: 10.1006/pmed.1998.0367. PMID 9922066